CLINICAL TRIAL: NCT07172685
Title: Exploratory Study on the Efficacy and Safety of Triple Therapy (ADT + Darolutamide + Docetaxel Chemotherapy) Combined With Transrectal High-Intensity Focused Ultrasound Focal Therapy in Metastatic Hormone-Sensitive Prostate Cancer (mHSPC) With High Tumor Burden
Brief Title: Study on Triple Therapy Combined With HIFU for High-Tumor-Burden mHSPC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSZ04
Record Dates: First submitted 2025-08-26; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-07

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — darolutamide; Docetaxel; Androgen Antagonists

STUDY DESIGN:
Intervention Model Description: This study is a single-arm prospective cohort study designed to evaluate the efficacy and safety of triple therapy (ADT + darolutamide + docetaxel) combined with transrectal high-intensity focused ultrasound (HIFU) focal therapy in patients with high-volume metastatic hormone-sensitive prostate cancer (mHSPC).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Arm (Experimental): The study plans to enroll 116 patients with high-volume metastatic hormone-sensitive prostate cancer (mHSPC) who will receive the following treatment regimen: Darolutamide , Docetaxel , ADT and transrectal high-intensity focused ultrasound (HIFU) focal therapy for the prostate. Patients will receive each drug according to the prescribing information, with dose adjustments based on adverse reactions (as per the prescribing guidelines).
  Interventions: Combination Product: Darolutamide , Docetaxel , ADT and Transrectal HIFU Focal Therapy

INTERVENTIONS:
Combination Product: Darolutamide , Docetaxel , ADT and Transrectal HIFU Focal Therapy — Darolutamide , Docetaxel , ADT and Transrectal HIFU Focal Therapy Group:
  Darolutamide (600 mg, orally, twice daily) GnRHa (Goserelin 10.8 mg sustained-release implant, subcutaneous injection, every 3 months) Docetaxel (75 mg/m², intravenous infusion, every 3 weeks, for 6 cycles) Dexamethasone (8 mg, orally, 12/3/1 hour before docetaxel infusion)* Prednisone/Prednisolone (at the investigator's discretion)* Transrectal High-Intensity Focused Ultrasound (HIFU) for prostate focal therapy (ablation extent determined based on MRI and biopsy findings; number of treatments ≤ 2)
  *Note: Dexamethasone and prednisone/prednisolone are adjunct medications and are not assigned as separate intervention arms; urinary catheter placement is a procedural detail and not listed as an intervention.

SUMMARY:
This study is a single-arm prospective cohort study designed to evaluate the efficacy and safety of triple therapy (ADT + darolutamide + docetaxel) combined with transrectal high-intensity focused ultrasound (HIFU) focal therapy in patients with high-tumor-burden metastatic hormone-sensitive prostate cancer (mHSPC).

A total of 116 high-tumor-burden mHSPC patients will be enrolled and are scheduled to receive the following treatment:

Darolutamide + Docetaxel + ADT + Transrectal HIFU Focal Therapy for the Prostate.

DETAILED DESCRIPTION:
Prostate cancer ranked as the second most commonly diagnosed cancer and the fifth leading cause of cancer death among men worldwide in 2020, with approximately 1.4 million new cases and 375,000 deaths. In China, both the incidence and mortality rates of prostate cancer have shown a significant upward trend.

For prostate cancer treatment, effective management of high-tumor-burden metastatic hormone-sensitive prostate cancer (mHSPC) is crucial for delaying disease progression and improving long-term survival, representing one of the most critical clinical challenges. Although androgen deprivation therapy (ADT) combined with docetaxel or novel hormonal therapy has been established as standard treatment in both domestic and international guidelines, the clinical adoption of these novel ADT-based combination regimens remains limited due to the risk of adverse events (AEs) associated with chemotherapy and prolonged hormone exposure.

Recent advances in mHSPC treatment have brought new hope. The phase III PEACE-1 trial demonstrated that adding abiraterone to standard ADT plus docetaxel significantly reduced mortality risk (median overall survival not reached vs. 4.4 years; HR, 0.75; 95% CI, 0.59-0.96; P=0.021).

SonaCare Medical's Sonablate HIFU system is a global leader in high-intensity focused ultrasound technology, being the first prostate tissue ablation device to receive FDA 510(k) clearance. On July 8, 2020, the Sonablate device obtained approval from China's National Medical Products Administration (NMPA Approval No. 20203010342) for treating both prostate cancer and benign prostatic hyperplasia.

Therefore, this project proposes a single-arm clinical study. From 2022 to 2025, eligible high-tumor-burden mHSPC patients will be enrolled after providing informed consent and baseline data collection. Participants will receive either:

* Apalutamide + docetaxel + ADT, or
* Apalutamide + ADT combined with transrectal high-intensity focused ultrasound (HIFU) focal therapy The primary endpoint is 3-year radiographic progression-free survival (rPFS) rate. Follow-up assessments will be conducted per protocol to evaluate efficacy and safety outcomes. This study aims to provide new therapeutic possibilities for high-tumor-burden mHSPC through combination therapy, potentially improving patient prognosis and reducing disease burden.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who agree to participate in the study and sign the informed consent form.
2. Age ≥18 years, male.
3. Histologically or cytologically confirmed prostate adenocarcinoma.
4. Bone scan, CT, or MRI showing ≥4 bone metastases (with ≥1 outside the pelvis or spine) or visceral metastases.
5. Newly diagnosed or recurrent disease after local therapy, with sensitivity to androgen deprivation therapy (ADT).
6. Patients who have received ADT (medical or surgical castration) with or without first-generation antiandrogens for ≤3 months, without evidence of soft tissue disease progression (per RECIST 1.1) or clinically significant PSA progression (≥50% increase from nadir with serum testosterone at castrate levels).
7. Planned treatment with docetaxel plus apalutamide and ADT, or apalutamide plus ADT.
8. ECOG Performance Status (PS) score of 0-1.
9. Adequate hematologic and organ function:

   * **Bone marrow function (without transfusion or growth factor support):**
   * Absolute neutrophil count (ANC) ≥1.5 × 10⁹/L (1500/μL)
   * Hemoglobin ≥90 g/L (9.0 g/dL)
   * Platelet count ≥100 × 10⁹/L (100,000/μL)
   * **Liver function:**
   * Total bilirubin (TBIL) ≤1.5 × ULN
   * AST, ALT, and alkaline phosphatase (ALP) ≤2.5 × ULN
   * **Renal function:**
   * Serum creatinine ≤1.5 × ULN **or** calculated creatinine clearance ≥30 mL/min (Cockcroft-Gault formula)
   * **Coagulation function (without anticoagulation therapy):** INR ≤1.5
10. Patients of reproductive potential must use effective contraception during the study and for 6 months after the last dose.

Exclusion Criteria:

1. Lesions located at the prostate apex or in areas inaccessible for focal therapy.
2. Beaded prostatic calculi or cysts >1 cm in diameter within the treatment or ultrasound pathway.
3. Urethral stricture or presence of metal/other implants in the urethra.
4. Prior rectal surgery.
5. History of or existing rectal fistula.
6. Rectal stenosis preventing transrectal ultrasound.
7. Rectal invasion.
8. Active severe urinary tract infection.
9. Severe cardiovascular or cerebrovascular disease affecting anesthesia/surgery.
10. History of hypersensitivity or intolerance to any study drugs.
11. Planned concurrent anticancer therapy during the study.
12. Prior treatment with second-generation androgen receptor (AR) inhibitors (e.g., apalutamide, enzalutamide, darolutamide), CYP17 inhibitors (e.g., abiraterone acetate, ketoconazole), chemotherapy, immunotherapy, or adjuvant/neoadjuvant therapy.
13. Use of herbal products with anti-prostate cancer or PSA-lowering effects (e.g., saw palmetto) within 4 weeks before study treatment.
14. History of seizures, medications that lower seizure threshold, or conditions predisposing to seizures within 12 months (including TIA, stroke, or traumatic brain injury with hospitalization).
15. Active cardiac disease within 6 months before treatment: severe/unstable angina, myocardial infarction, congestive heart failure (NYHA Class III/IV), or arrhythmia requiring medication.
16. Conditions impairing drug absorption (e.g., dysphagia, chronic diarrhea, intestinal obstruction).
17. Immunodeficiency (e.g., HIV-positive, congenital/acquired immunodeficiency) or organ transplant history.
18. Known brain metastases.
19. Other malignancies within 5 years (except cured basal cell carcinoma or cervical carcinoma in situ).
20. Concurrent participation in another investigational drug/device trial.
21. Poor compliance likely to hinder treatment/follow-up.
22. Uncontrolled comorbidities (e.g., hypertension, diabetes, neuropsychiatric disorders) that may compromise safety or confound results, per investigator judgment.
23. Any other condition deemed unsuitable for inclusion by the investigator.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2025-07-30 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
PSA Evaluation | PSA Response Rate at Week 12
  Time to PSA Progression

SECONDARY OUTCOMES:
PFS | Time from randomization to tumor progression (any aspect) or death (any cause), or until a maximum of 2 years of drug exposure per subject, whichever occurs first.
PSA ≤0.2 ng/ml Response Rate | Months 3, 6, and 12
PSA50 and PSA90 Response Rates | Month 6

CONTACTS AND LOCATIONS:
Overall Officials: Shouzhen Chen, Dr., Study Chair — Qilu Hospital of Shandong University
Locations (1):
- Qilu hospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Morris MJ, Rathkopf DE, Novotny W, Gibbons JA, Peterson AC, Khondker Z, Ouatas T, Scher HI, Fleming MT. Phase Ib Study of Enzalutamide in Combination with Docetaxel in Men with Metastatic Castration-Resistant Prostate Cancer. Clin Cancer Res. 2016 Aug 1;22(15):3774-81. doi: 10.1158/1078-0432.CCR-15-2638. Epub 2016 Feb 8. PMID 26858312
- [Background] Gan L, Chen S, Wang Y, Watahiki A, Bohrer L, Sun Z, Wang Y, Huang H. Inhibition of the androgen receptor as a novel mechanism of taxol chemotherapy in prostate cancer. Cancer Res. 2009 Nov 1;69(21):8386-94. doi: 10.1158/0008-5472.CAN-09-1504. Epub 2009 Oct 13. PMID 19826044
- [Background] Darshan MS, Loftus MS, Thadani-Mulero M, Levy BP, Escuin D, Zhou XK, Gjyrezi A, Chanel-Vos C, Shen R, Tagawa ST, Bander NH, Nanus DM, Giannakakou P. Taxane-induced blockade to nuclear accumulation of the androgen receptor predicts clinical responses in metastatic prostate cancer. Cancer Res. 2011 Sep 15;71(18):6019-29. doi: 10.1158/0008-5472.CAN-11-1417. Epub 2011 Jul 28. PMID 21799031
- [Background] Zhu Y, Liu C, Armstrong C, Lou W, Sandher A, Gao AC. Antiandrogens Inhibit ABCB1 Efflux and ATPase Activity and Reverse Docetaxel Resistance in Advanced Prostate Cancer. Clin Cancer Res. 2015 Sep 15;21(18):4133-42. doi: 10.1158/1078-0432.CCR-15-0269. Epub 2015 May 20. PMID 25995342
- [Background] Galletti G, Matov A, Beltran H, Fontugne J, Miguel Mosquera J, Cheung C, MacDonald TY, Sung M, O'Toole S, Kench JG, Suk Chae S, Kimovski D, Tagawa ST, Nanus DM, Rubin MA, Horvath LG, Giannakakou P, Rickman DS. ERG induces taxane resistance in castration-resistant prostate cancer. Nat Commun. 2014 Nov 25;5:5548. doi: 10.1038/ncomms6548. PMID 25420520
- [Background] Eigl BJ, Eggener SE, Baybik J, Ettinger S, Chi KN, Nelson C, Wang Z, Gleave ME. Timing is everything: preclinical evidence supporting simultaneous rather than sequential chemohormonal therapy for prostate cancer. Clin Cancer Res. 2005 Jul 1;11(13):4905-11. doi: 10.1158/1078-0432.CCR-04-2140. PMID 16000589
- [Background] Ueda Y, Matsubara N, Takizawa I, Nishiyama T, Tabata K, Satoh T, Kamiya N, Suzuki H, Kawahara T, Uemura H. A multicenter retrospective analysis of sequential treatment of abiraterone acetate followed by docetaxel in Japanese patients with metastatic castration-resistant prostate cancer. Jpn J Clin Oncol. 2015 Aug;45(8):774-9. doi: 10.1093/jjco/hyv070. Epub 2015 May 15. PMID 25981621
- [Background] Zhang T, Dhawan MS, Healy P, George DJ, Harrison MR, Oldan J, Chin B, Armstrong AJ. Exploring the Clinical Benefit of Docetaxel or Enzalutamide After Disease Progression During Abiraterone Acetate and Prednisone Treatment in Men With Metastatic Castration-Resistant Prostate Cancer. Clin Genitourin Cancer. 2015 Aug;13(4):392-399. doi: 10.1016/j.clgc.2015.01.004. Epub 2015 Jan 24. PMID 25708161
- [Background] Mezynski J, Pezaro C, Bianchini D, Zivi A, Sandhu S, Thompson E, Hunt J, Sheridan E, Baikady B, Sarvadikar A, Maier G, Reid AHM, Mulick Cassidy A, Olmos D, Attard G, de Bono J. Antitumour activity of docetaxel following treatment with the CYP17A1 inhibitor abiraterone: clinical evidence for cross-resistance? Ann Oncol. 2012 Nov;23(11):2943-2947. doi: 10.1093/annonc/mds119. Epub 2012 Jul 5. PMID 22771826
- [Background] de Bono JS, Chowdhury S, Feyerabend S, Elliott T, Grande E, Melhem-Bertrandt A, Baron B, Hirmand M, Werbrouck P, Fizazi K. Antitumour Activity and Safety of Enzalutamide in Patients with Metastatic Castration-resistant Prostate Cancer Previously Treated with Abiraterone Acetate Plus Prednisone for >/=24 weeks in Europe. Eur Urol. 2018 Jul;74(1):37-45. doi: 10.1016/j.eururo.2017.07.035. Epub 2017 Aug 23. PMID 28844372
- [Background] Matsubara N, Yamada Y, Tabata KI, Satoh T, Kamiya N, Suzuki H, Kawahara T, Uemura H, Yano A, Kawakami S, Otsuka M, Fukasawa S. Abiraterone Followed by Enzalutamide Versus Enzalutamide Followed by Abiraterone in Chemotherapy-naive Patients With Metastatic Castration-resistant Prostate Cancer. Clin Genitourin Cancer. 2018 Apr;16(2):142-148. doi: 10.1016/j.clgc.2017.09.008. Epub 2017 Sep 23. PMID 29042308
- [Background] Khalaf DJ, Annala M, Taavitsainen S, Finch DL, Oja C, Vergidis J, Zulfiqar M, Sunderland K, Azad AA, Kollmannsberger CK, Eigl BJ, Noonan K, Wadhwa D, Attwell A, Keith B, Ellard SL, Le L, Gleave ME, Wyatt AW, Chi KN. Optimal sequencing of enzalutamide and abiraterone acetate plus prednisone in metastatic castration-resistant prostate cancer: a multicentre, randomised, open-label, phase 2, crossover trial. Lancet Oncol. 2019 Dec;20(12):1730-1739. doi: 10.1016/S1470-2045(19)30688-6. Epub 2019 Nov 11. PMID 31727538
- [Background] McGuire S. World Cancer Report 2014. Geneva, Switzerland: World Health Organization, International Agency for Research on Cancer, WHO Press, 2015. Adv Nutr. 2016 Mar 15;7(2):418-9. doi: 10.3945/an.116.012211. Print 2016 Mar. No abstract available. PMID 26980827